CLINICAL TRIAL: NCT05588622
Title: Feasibility of a Therapist-Supported Digital Mental Health Intervention in Addressing Mental Health Symptoms Among People With Cancer: A Mixed Methods Study
Brief Title: Meru Health Program for Cancer Patients With Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meru Health, Inc. (Industry)
Collaborators: Cancer Support Community, Headquarters (Other); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Nicholas Peiper, PhD, MPH, Director of Research, Meru Health, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-MERU-117
Record Dates: First submitted 2022-10-13; First posted 2022-10-20 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Depression; Anxiety
Keywords: Mental Health; Digital Mental Health; Depression; Anxiety; Meru Health
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): This single-arm study will enroll all 20 participants in the Meru Health Program.
  Interventions: Behavioral: Meru Health Program

INTERVENTIONS:
Behavioral: Meru Health Program — The Meru Health Program is a 12-week, evidence-based, smartphone-delivered, therapist-supported digital mental health intervention with as-needed psychiatrist oversight. Enrolled participants work through the program with a cohort of peers similarly affected by depression, with whom they can engage in confidential, anonymous, voluntary group chats overseen by a licensed clinical therapist. The MHP incorporates a continuous care model including daily interaction with a dedicated clinician, several evidence-based treatment components such as cognitive behavioral therapy (CBT), behavioral activation therapy, and mindfulness meditation (MM), as well as promising newer types of depression treatments such as HRVB, nutritional psychiatry, and sleep training. Practices are introduced to weekly topics via video lessons that are reinforced via CBT practices, meditations, and biofeedback sessions and therapist messaging.

SUMMARY:
The primary objective of this study is to evaluate clinical outcomes among people with cancer who participate in a 12-week therapist-supported digital mental health intervention (DMHI) called the Meru Health Program (MHP). Study participants (N=20) will be referred to the MHP through the Cancer Support Community (CSC) Helpline and network of Gilda's Club locations. The main outcomes will be depression symptoms, anxiety symptoms, health-related quality of life (HRQoL), intervention adherence, and intervention satisfaction. The secondary objective will be to determine the acceptability of the screening and referral process from the CSC networks into the MHP. Data pertaining to implementability will be collected from study participants, MHP clinicians, and CSC staff.

DETAILED DESCRIPTION:
The goal of this single-arm intervention study is to test the feasibility of the Meru Health Program (MHP) in reducing symptoms of depression and anxiety among 20 people with cancer referred from the Cancer Support Community (CSC). The MHP is a 12-week digital mental health intervention delivered via a smartphone app. The intervention focuses on cognitive behavioral techniques and mindfulness skills with the aim of improving mental health symptoms. The platform provides informational videos, skills practices, group discussion, and messaging with a licensed clinician employed by Meru Health. The licensed clinician supports patients as needed and reviews engagement logs within the app. As part of the intervention, depression and anxiety symptoms are measured on a biweekly basis over 12 weeks. For this study, self-reported surveys will be administered at baseline, week 12, and 2-months post-treatment to measure health-related quality of life and intervention satisfaction. In-depth interviews will be conducted with patients. Two focus groups will be conducted with MHP clinicians and CSC navigators to understand barriers and facilitators to the screening processes and intervention delivery.

ELIGIBILITY:
Inclusion Criteria:

* Positive screen (score >= 3 out of 8) on the anxiety or depression subscale of the CSS 15+ Questionnaire
* PHQ-9 and/or GAD-7 score >= 5 at clinical intake
* Willing to commit to the Meru Health Program if selected
* Proficient in the English language
* At least 18 years of age at the time of enrollment
* Has a valid mailing address
* Owns 1 of the 3 past versions of an Apple or Android mobile phone operating system
* Currently in active cancer treatment at the time of enrollment

Exclusion Criteria:

* Active suicide intent with plan to act
* Substance use disorder in the past 3 months
* Lifetime bipolar disorder
* Lifetime psychotic disorder
* Currently pregnant
* Less than 3 months postpartum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change in PHQ-9 Scores | Baseline, Week 12, and 2 Month Follow-Up time points
  9-item questionnaire to measure depression symptoms
Change in GAD-7 Scores | Baseline, Week 12, and 2 Month Follow-Up time points
  7-item questionnaire to measure anxiety symptoms
Change in Eurohis-QOL-8 Scores | Baseline, Week 12, and 2 Month Follow-Up time points
  8-item Quality of Life questionnaire.
Change in CSS 15+ Scores | Baseline and Week 12 time points
  15-item questionnaire to measure psychological distress experiencing and receiving treatment for cancer.

SECONDARY OUTCOMES:
Change in Burnout Scores | Baseline, Week 12, and 2 Month Follow-Up
  A single-item questionnaire to address worker stress and burnout.

CONTACTS AND LOCATIONS:
Locations (1):
- Online Digital Mental Health Clinic, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No